CLINICAL TRIAL: NCT00003400
Title: High Dose Chemotherapy With Stem Cell Rescue Followed By Consolidation Treatment in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MSGCC-9748; CDR0000066404 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1436
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Filgrastim; Carmustine; Cisplatin; Melphalan; Vinorelbine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cisplatin
Drug: melphalan
Drug: vinorelbine tartrate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high dose chemotherapy plus peripheral stem cell transplantation followed by combination chemotherapy in treating patients with metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete and partial remission rates and event free and overall survival of patients with metastatic hormone refractory prostate cancer treated with high dose chemotherapy plus peripheral stem cell transplantation followed by consolidation chemotherapy. II. Evaluate the toxic effects associated with this treatment in these patients. III. Evaluate the quality of life, and need for analgesics, in these patients.

OUTLINE: Patients are stratified by stage of disease and extent of metastatic disease. Patients receive daily filgrastim (G-CSF) subcutaneously for 4 days until peripheral blood stem cells are collected. Patients then receive carmustine IV over 2 hours on day -2 and melphalan IV over 20 minutes on day -1. Stem cell infusion will be on day 0. At 3, 6, 9, and 12 months after transplant, patients receive vinorelbine IV over 10 minutes and cisplatin IV over 24 hours. Quality of life and pain are assessed before the transplantation, just before discharge after transplantation, prior to each consolidation course, and then at 3, 6, and 12 months after the final course of chemotherapy. Patients are followed at least every 3 months for the first 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 18-45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic hormone refractory adenocarcinoma of the prostate that is progressive on hormone based therapy, as demonstrated by: New metastatic lesion Consecutive series of increasing PSA levels following hormonal therapy No CNS disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: SWOG 0-2 (unless due to bone pain) Life expectancy: Not specified Hematopoietic: CD34+ at least 4 million/kg Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal No active chronic hepatitis or liver cirrhosis Renal: Creatinine no greater than 3 mg/dL Cardiovascular: Left ventricular ejection fraction at least 50% Pulmonary: FVC, FEV1, and corrected DLCO at least 50% of predicted (high resolution CT scan of chest and P02 at least 70 if unable to complete PFTs) Other: No active infection requiring intravenous antibiotics Not HIV positive

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than one course of cytotoxic chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1998-09 (Actual); Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido J. Tricot, MD, PhD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States